CLINICAL TRIAL: NCT02877394
Title: Use of a Squatting Assist Device in Patients With Constipation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adil Bharucha, MBBS, MD, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-004548
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Squatting Assist Device (Experimental): The Squatty Potty is a 7 inch tall stool to assist subjects in maintaining a squatting position while using a toilet. While sitting on the toilet, the subject supports her feet on the Squatty Potty.
  Interventions: Device: Squatting Assist Device
- Sham Squatting Assist Device (Sham Comparator): This stool will be 2 inches tall and be similar in appearance to the Squatty Potty. While sitting on the toilet, the subject supports her feet on the 2 inch high stool.
  Interventions: Device: Sham Squatting Assist Device

INTERVENTIONS:
Device: Squatting Assist Device — The Squatty Potty is a 7 inch tall stool to assist subjects in maintaining a squatting position while using a toilet. While sitting on the toilet, the subject supports her feet on the Squatty Potty.
  Other Names: Squatty Potty
  Arms: Squatting Assist Device
Device: Sham Squatting Assist Device — This stool will be 2 inches tall and be similar in appearance to the Squatty Potty. While sitting on the toilet, the subject supports her feet on the 2 inch high stool.
  Arms: Sham Squatting Assist Device

SUMMARY:
Constipation is a very common problem. Western style toilets that are nearly universal in the United States require the person to sit on the toilet. However, results from uncontrolled studies suggests that a squatting posture (as prevalent in many foreign countries) may be better at facilitating evacuation compared to a Western style commode. One uncontrolled, unpublished study suggests that a footstool improved bowel symptoms in nearly 98% of 153 constipated participants. Hence, the investigators propose to evaluate the benefits of a footstool on symptoms and anorectal functions in constipated patients. Hypothesis: the regular squatting assist device (7 inches) but not a sham device (2 inches tall) will improve symptoms of constipation.

ELIGIBILITY:
Inclusion criteria:

* Able to communicate adequately with the investigator and to comply with the requirements for the entire study
* Meet Rome III criteria for functional constipation as assessed by questionnaires in period 1, i.e., report at least 2 of the following symptoms for last 3 months or more with symptom onset at least 6 months prior to diagnosis: a) <3 SBMs/week b) hard or lumpy stools ≥ 25% of time c) straining ≥ 25% of time d) sense of incomplete evacuation ≥ 25% of time e) feeling of anorectal blockage ≥ 25% of time or f) manual maneuvers to facilitate defecation ≥ 25% of time. Patients who meet Rome III criteria for irritable bowel syndrome will also be eligible provided they also meet above criteria.

Exclusion criteria:

* Current use of opioid analgesics. Patients on opioids will be allowed to participate if they have discontinued them for at least 3 days (72 hrs.) before date of screening and are willing to stay off them for the duration of the study.
* Current use of anticholinergics (e.g. nortriptyline, amitriptyline, hyoscyamine). Patients who use low dose tricyclic antidepressants (nortriptyline upto 50 mg/day or amitriptyline upto 25 mg/day ) will be eligible provided they do not increase the dose during the study period. Patients on higher doses or on other anticholinergics are eligible to participate if they can discontinue their medication at least 3 days (72 hrs) before the date of screening and are willing to stay off them till the study is complete.
* Current use of laxatives (MiraLax, Ex-lax, senna, herbal supplements), linaclotide, lubiprostone, and prucalopride to treat constipation- patients using these medications will be eligible to participate if they can discontinue the medication at least 3 days (72 hrs.) before the date of screening and are willing to stay off them till the study is complete.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Weekly Complete Spontaneous Bowel Movement (CSBM) Frequency | baseline, 4 weeks
  Weekly CSBM Frequency = (Number of CSBMs recorded in 7 days/Number of days with bowel entries in subject diary) X 7

CONTACTS AND LOCATIONS:
Overall Officials: Adil E Bharucha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No